CLINICAL TRIAL: NCT05873595
Title: Clinical Understanding Through Real-world Data to Validate Effectiveness of Treatments in Peyronie's Disease
Brief Title: Real-World Data Study to Understand Effectiveness of Treatments in Peyronie's Disease
Acronym: CURVE-PD
Status: Terminated | Type: Observational
Why Stopped: Endo determined to discontinue its registries and the CURVE registry enrollment has been closed.
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: EP02REG
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Peyronie's Disease
Keywords: Real world data; Retrospective; Prospective; Registry
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

SUMMARY:
This is an observational study, meaning participants will not receive any investigational treatment as part of this study.

Researchers will collect real-world data (RWD) to gain a more in-depth knowledge of the treatment of Peyronie's Disease (PD) to evaluate the management of PD.

DETAILED DESCRIPTION:
Each participant of the study will have their data collected from the date of confirmed diagnosis of PD to the date of enrollment in the registry, post consent. Data will be collected from the participant's clinical records as well as from the participant directly. Data will be collected through Pulse Infoframe's technology platform.

ELIGIBILITY:
Key Inclusion Criteria:

* Any adult with a confirmed clinical diagnosis of PD.
* Age 18 years (or age of majority in their jurisdiction) or older at time of enrollment.
* Willing to participate in the registry (including completion of ePROs) and complete the informed consent form.
* Having received PD treatment within 2 weeks before enrollment, at enrollment or any time after the date of enrollment. After a confirmed diagnosis of PD, not having received PD treatment.
* Able to participate in English based registry.

Key Exclusion criteria:

* Not having a clinical diagnosis of PD.
* Age less than 18 years.
* Do not provide informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a confirmed diagnosis of PD will be enrolled in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants Receiving Each Treatment Type for PD | Up to 12 months

SECONDARY OUTCOMES:
Change from Baseline in Peyronie's Disease Questionnaire (PDQ) Score | Up to 12 months
Change from Baseline in International Index of Erectile Function (IIEF) Score | Up to 12 months
Change from Baseline in Patient Health Questionnaire-9 (PHQ-9) Score | Up to 12 months
Change from Baseline in Beck Anxiety Inventory (BAI) Scale Score | Up to 12 months
Participant Satisfaction Questionnaire | Up to 12 months
Number of Participants Receiving Post-Procedural Care by the Treating Physician | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Endo Pharmaceuticals
Locations (7):
- United States (7):
  - Endo Pharmaceuticals Clinical Site 2, San Diego, California
  - Endo Pharmaceuticals Clinical Site 3, Miami, Florida
  - Endo Pharmaceuticals Clinical Site 6, Greenwood, Indiana
  - Endo Pharmaceuticals Clinical Site 5, Lansing, Michigan
  - Endo Pharmaceuticals Clinical Site 7, Gahanna, Ohio
  - Endo Pharmaceuticals Clinical Site 4, Houston, Texas
  - Endo Pharmaceuticals Clinical Site 1, Orem, Utah